CLINICAL TRIAL: NCT01286753
Title: An Open-Label, Multi-Center Phase II Study of the BRAF Inhibitor Vemurafenib in Patients With Metastatic or Unresectable Papillary Thyroid Cancer (PTC) Positive for the BRAF V600 Mutation and Resistant to Radioactive Iodine
Brief Title: A Study of Vemurafenib (RO5185426) in Participants With Metastatic or Unresectable Papillary Thyroid Cancer Positive for the BRAF V600 Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO25530; 2010-024133-23
Record Dates: First submitted 2011-01-28; First posted 2011-01-31 (Estimated); Results first posted 2016-09-07 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tyrosine Kinase Inhibitor (TKI) Naive (Experimental): Vemurafenib in participants naive to any prior systemic TKI therapy.
  Interventions: Drug: Vemurafenib
- TKI Experienced (Experimental): Vemurafenib in participants previously treated with TKI therapy active against vascular endothelial growth factor receptor 2 (VEGFR).
  Interventions: Drug: Vemurafenib

INTERVENTIONS:
Drug: Vemurafenib — Vemurafenib 960 mg orally twice daily.
  Other Names: Zelboraf®; RO5185426

SUMMARY:
This open-label, multi-center study will evaluate the safety and efficacy of Vemurafenib (RO5185426) in participants with metastatic or unresectable papillary thyroid cancer (PTC) positive for the BRAF V600 mutation and resistant to radioactive iodine therapy. Participants will receive vemurafenib 960 milligrams (mg) orally twice daily until progressive disease or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants. >/= 18 years of age
* Histologically confirmed metastatic or unresectable papillary thyroid cancer for which standard curative or palliative measures do not exist or are no longer effective; participants whose tumors exhibit areas of "other histology" may be enrolled, provided the tumor histology remains predominantly papillary
* Positive for BRAF V600 mutation (Roche Cobas 4800 BRAF V600 Mutation Test)
* Radioactive Iodine resistant disease
* Prior therapy excluding (Cohort 1, TKI Naive) or including (Cohort 2, TKI Experienced) TKI
* Clinically relevant disease progression according to RECIST criteria within the prior 14 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate hematological, renal and liver function

Exclusion Criteria:

* Histological diagnosis other than papillary PTC, including squamous cell variants of PTC or PTC with areas of squamous metaplasia
* Active or untreated central nervous system metastases
* History of or known carcinomatous meningitis
* Anticipated or ongoing administration of any anti-cancer therapies other than those administered in the study
* Active squamous cell skin cancer that has not been excised or adequately healed post excision
* Previous treatment with any agent that specifically and selectively targets the MEK or BRAF pathway
* Prior radiotherapy to the only measurable lesion
* Clinically relevant cardio-vascular disease or event within the prior 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-06; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- United States (8):
  - Torrance, California
  - New Haven, Connecticut
  - Chicago, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - New York, New York
  - Philadelphia, Pennsylvania
  - Houston, Texas
- France (3):
  - Lyon
  - Paris
  - Villejuif
- Italy (2):
  - Milan, Lombardy
  - Pisa, Tuscany
- Netherlands (2):
  - Groningen
  - Leiden

REFERENCES:
- [Derived] Brose MS, Cabanillas ME, Cohen EE, Wirth LJ, Riehl T, Yue H, Sherman SI, Sherman EJ. Vemurafenib in patients with BRAF(V600E)-positive metastatic or unresectable papillary thyroid cancer refractory to radioactive iodine: a non-randomised, multicentre, open-label, phase 2 trial. Lancet Oncol. 2016 Sep;17(9):1272-82. doi: 10.1016/S1470-2045(16)30166-8. Epub 2016 Jul 23. PMID 27460442

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Written informed consent for participation in the study was obtained before performing any study-specific screening tests or evaluations.
Groups:
- Tyrosine Kinase Inhibitor (TKI) Naive: Vemurafenib 960 milligrams (mg) orally twice daily in participants naive to any prior systemic TKI therapy.
- TKI Experienced: Vemurafenib 960 mg orally twice daily in participants previously treated with TKI therapy active against vascular endothelial growth factor receptor 2 (VEGFR).
Period: Overall Study
Arm/Group | Tyrosine Kinase Inhibitor (TKI) Naive | TKI Experienced
Started | 26 | 25
Completed | 0 | 0
Not Completed | 26 | 25
Not completed — Adverse Event | 7 | 6
Not completed — Progression | 11 | 13
Not completed — Refused Treatment | 1 | 0
Not completed — Withdrawal of Consent | 0 | 2
Not completed — Discontinued to Join Extension Study | 6 | 4
Not completed — Participant to Receive Radiotherapy | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population, defined as all enrolled participants.
Groups:
- TKI Naive: Vemurafenib 960 mg orally twice daily in participants naive to any prior systemic TKI therapy.
- TKI Experienced: Vemurafenib 960 mg orally twice daily in participants previously treated with TKI therapy active against VEGFR.
- Total: Total of all reporting groups
Arm/Group | TKI Naive | TKI Experienced | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (13.5) | 65.2 (9.1) | 64.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate in TKI-Naive Participants
Description: Best overall response rate was assessed by the investigators according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Best overall response rate: the percentage of participants with best objective response of complete response (CR) or partial response (PR) (calculated as the number of participants with best response CR or PR divided by the total number of efficacy-evaluable participants). CR: disappearance of all target lesions with reduction in target/non-target pathological lymph nodes to < 10 millimeters (mm). PR: ≥ 30% decrease in the sum of diameters of target lesions, compared to the baseline sum diameters.
Time Frame: Up to approximately 4 years
Population: Efficacy population (TKI Naive group only), defined as all enrolled participants who received at least one dose of study treatment and excluding 3 participants in the TKI Experienced group who had previous BRAFi or MEKi treatment or withdrew consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TKI Naive
Number analyzed (Participants) | 26
percentage of participants | 42.3 [23.35 to 63.08]

2. Secondary Outcome: Best Overall Response Rate in TKI-Experienced Participants
Description: Best overall response rate was assessed by the investigators according to RECIST v1.1. Best overall response rate: the percentage of participants with best objective response of CR or PR (calculated as the number of participants with best response CR or PR divided by the total number of efficacy-evaluable participants). CR: disappearance of all target lesions with reduction in target/non-target pathological lymph nodes to < 10 mm. PR: ≥ 30% decrease in the sum of diameters of target lesions, compared to the baseline sum diameters.
Time Frame: Up to approximately 4 years
Population: Efficacy population (TKI Experienced group only), defined as all enrolled participants who received at least one dose of study treatment and excluding 3 participants in the TKI Experienced group who had previous BRAFi or MEKi treatment or withdrew consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TKI Experienced
Number analyzed (Participants) | 22
percentage of participants | 27.3 [10.73 to 50.22]

3. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate: the percentage of participants with confirmed CR, PR, or stable disease (SD; maintained for at least 6 months) as assessed by investigators according to RECIST v1.1. CR: disappearance of all target lesions with reduction in target/non-target pathological lymph nodes to < 10 mm. PR: ≥ 30% decrease in the sum of diameters of target lesions, compared to the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, compared to the baseline sum diameters.
Time Frame: Up to approximately 4 years
Population: Efficacy population, defined as all enrolled participants who received at least one dose of study treatment and excluding 3 participants in the TKI Experienced group who had previous BRAFi or MEKi treatment or withdrew consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TKI Naive | TKI Experienced
Number analyzed (Participants) | 26 | 22
percentage of participants | 73.1 [52.21 to 88.43] | 54.5 [32.21 to 75.61]

4. Secondary Outcome: Duration of Response
Description: Duration of response (for participants with confirmed best response CR or PR): the interval between earliest qualifying response and date of progression of disease (PD) or death for any cause, whichever occurred first; participants with no documented progression after CR or PR were censored at the date of last known CR or PR, respectively. CR: disappearance of all target lesions with reduction in target/non-target pathological lymph nodes to < 10 mm. PR: ≥ 30% decrease in the sum of diameters of target lesions, compared to the baseline sum diameters. PD: ≥ 20% increase in the sum of diameters of target lesions, compared to the smallest sum on study.
Time Frame: From the date of first qualifying response to the date of PD or death for any cause (up to approximately 4 years)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TKI Naive | TKI Experienced
Number analyzed (Participants) | 26 | 22
months | 9.5 [5.7 to NA] — NA = Not estimable due to an insufficient number of events. | 7.4 [3.7 to NA] — NA = Not estimable due to an insufficient number of events.

5. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival: the interval between the day of first treatment and the first documentation of PD or death; participants who were withdrawn from the study without documented progression were censored at the date of the last tumor assessment when the participant was known to be progression-free; participants without post baseline tumor assessments were censored at the time of enrollment. PD: ≥ 20% increase in the sum of diameters of target lesions, compared to the smallest sum on study.
Time Frame: From the day of first treatment until the first documented PD or death (up to approximately 4 years)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TKI Naive | TKI Experienced
Number analyzed (Participants) | 26 | 22
months | 18.2 [15.5 to 29.3] | 8.9 [5.5 to 27.7]

6. Secondary Outcome: Overall Survival
Description: Overall survival: the interval between the date of first treatment to the date of death, regardless of the cause of death; participants who were alive at the time of the analysis were censored at the date of the last known alive; participants with no post baseline information were censored at the time of enrollment.
Time Frame: From the date of first treatment to the date of death for any cause (up to approximately 4 years)
Population: Intent-to-Treat population, defined as all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TKI Naive | TKI Experienced
Number analyzed (Participants) | 26 | 25
months | NA [28.3 to NA] — NA = Not estimable due to an insufficient number of events. | 14.4 [8.2 to 29.1]

7. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Baseline until 28 days after the last dose of study treatment or until initiation of another anti-cancer therapy, whichever occurred first (up to approximately 4 years)
Population: Safety population, defined as enrolled participants who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | TKI Naive | TKI Experienced
Number analyzed (Participants) | 26 | 25
percentage of participants | 100 | 100

8. Secondary Outcome: Pharmacokinetics of Vemurafenib: Area Under the Concentration-Time Curve (AUC)
Description: AUC is a measure of the drug or biologic concentration in the body following administration.
Time Frame: Up to approximately 4 years
Population: Data were not collected for this outcome.
Arm/Group | TKI Naive | TKI Experienced
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline until 28 days after the last dose of study treatment or until initiation of another anti-cancer therapy, whichever occurred first (up to approximately 4 years)
Description: Safety population, defined as enrolled participants who received at least one dose of study treatment.
Arm/Group | TKI Naive | TKI Experienced
Serious Adverse Events (participants affected / at risk) | 16/26 | 18/25
Other Adverse Events (participants affected / at risk) | 26/26 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TKI Naive (N=26) | TKI Experienced (N=25)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 5
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Large intestinal perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oral lichen planus (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Larygeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Viral labyrinthitis (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Seizure (Nervous system disorders) | 0 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesions (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TKI Naive (N=26) | TKI Experienced (N=25)
Anaemia (Blood and lymphatic system disorders) | 9 | 13
Leukopenia (Blood and lymphatic system disorders) | 3 | 1
Lymphopenia (Blood and lymphatic system disorders) | 5 | 5
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Cataract (Eye disorders) | 2 | 0
Photophobia (Eye disorders) | 3 | 1
Scleral discolouration (Eye disorders) | 1 | 2
Vision blurred (Eye disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 12 | 6
Dry mouth (Gastrointestinal disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 4 | 3
Gingival bleeding (Gastrointestinal disorders) | 2 | 0
Leukoplakia oral (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 13 | 7
Oral disorder (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 6 | 6
Asthenia (General disorders) | 5 | 3
Chills (General disorders) | 2 | 4
Cyst (General disorders) | 5 | 0
Fatigue (General disorders) | 18 | 14
Induration (General disorders) | 2 | 0
Localised oedema (General disorders) | 2 | 0
Nodule (General disorders) | 3 | 1
Oedema peripheral (General disorders) | 4 | 7
Peripheral swelling (General disorders) | 0 | 3
Pyrexia (General disorders) | 1 | 6
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1
Bronchitis (Infections and infestations) | 3 | 2
Conjunctivitis (Infections and infestations) | 4 | 1
Folliculitis (Infections and infestations) | 2 | 1
Hordeolum (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 3 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2
Oral candidiasis (Infections and infestations) | 3 | 2
Rhinitis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 2 | 0
Skin infection (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 3 | 4
Fall (Injury, poisoning and procedural complications) | 2 | 1
Sunburn (Injury, poisoning and procedural complications) | 3 | 4
Alanine aminotransferase increased (Investigations) | 4 | 5
Aspartate aminotransferase increased (Investigations) | 5 | 6
Blood alkaline phosphatase increased (Investigations) | 7 | 6
Blood bilirubin increased (Investigations) | 10 | 10
Blood creatinine increased (Investigations) | 13 | 6
Blood glucose increased (Investigations) | 2 | 0
Blood pressure increased (Investigations) | 0 | 2
Blood thyroid stimulating hormone increased (Investigations) | 2 | 1
Blood uric acid increased (Investigations) | 4 | 2
Electrocardiogram QT prolonged (Investigations) | 4 | 0
Gamma-glutamyltransferase increased (Investigations) | 7 | 7
Haemoglobin decreased (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 0 | 2
Weight decreased (Investigations) | 14 | 14
White blood cell count decreased (Investigations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 13 | 11
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 7
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 8
Dizziness (Nervous system disorders) | 2 | 8
Dysgeusia (Nervous system disorders) | 14 | 6
Headache (Nervous system disorders) | 7 | 6
Paraesthesia (Nervous system disorders) | 6 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2
Agitation (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 4 | 3
Haematuria (Renal and urinary disorders) | 2 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 7 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 7
Dermal cyst (Skin and subcutaneous tissue disorders) | 4 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 6
Erythema (Skin and subcutaneous tissue disorders) | 2 | 5
Erythema nodosum (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 11 | 6
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 4 | 3
Macule (Skin and subcutaneous tissue disorders) | 2 | 0
Milia (Skin and subcutaneous tissue disorders) | 2 | 0
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 | 6
Panniculitis (Skin and subcutaneous tissue disorders) | 2 | 1
Papule (Skin and subcutaneous tissue disorders) | 2 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 8 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 11 | 7
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 3 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 5 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 5 | 4
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 2
Hypertension (Vascular disorders) | 6 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.